CLINICAL TRIAL: NCT00577681
Title: Lipoproteins, HIV, and Antiretroviral Therapy in SMART
Brief Title: Understanding the Increased Risk of Cardiovascular Disease in People With HIV
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0708M14181; R01HL090934 (NIH); R01HL090934-01 (NIH)
Record Dates: First submitted 2007-12-17; First posted 2007-12-20 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: HIV Infections
Keywords: HIV; Lipoproteins; Inflammatory Markers; Coagulation Markers; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The plasma specimens will be collected using EDTA plasma tubes. For each specimen, four transport tubes (Sarstedt 2.0 mL Micro Tube), each containing 1 mL of plasma, will be prepared and labeled with preprinted bar coded labels. The preprinted bar coded labels specify the patient identification code (PID), visit and specimen type, and the protocol and vial ID. Specimens will be frozen at negative 70 degrees Celcius and shipped on dry ice to a central repository, Advanced Biomedical Laboratories, Cinnaminson, New Jersey, where they will be scanned and put into storage. Paperwork documenting the specimens will be processed by the SDMC, and electronic files will be sent to the central repository.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Participants from the SMART study who were randomly assigned to episodic or continuous ART and who have no history of CVD
  Interventions: Drug: Antiretroviral Therapy (ART)
- 2: Participants from the SMART study who were randomly assigned to episodic or continuous ART and who experienced a major CVD event during the study, analyzed along with 2 matched controls
  Interventions: Drug: Antiretroviral Therapy (ART)
- 3: Participants from the SMART study who have no previous use of ART or have taken ART but not done so within 6 months prior to study entry; allows for a comparison of immediate ART versus deferred ART
  Interventions: Drug: Antiretroviral Therapy (ART)

INTERVENTIONS:
Drug: Antiretroviral Therapy (ART) — Either episodic ART or continuous ART. All groups will have plasma specimens taken to compare changes in lipoprotein particle sizes and numbers and changes in inflammatory and coagulation markers.
  Other Names: Anti-HIV therapy

SUMMARY:
HIV is a virus that can lead to acquired immunodeficiency syndrome (AIDS), a disease for which there is not yet a cure. Antiretroviral therapy (ART) has proven an effective treatment for inhibiting the replication of HIV, allowing for improved quality of life and survival. Previous studies indicate that episodic use of ART is associated with increased risk of cardiovascular disease (CVD). This study will determine mechanisms underlying the increased CVD risk among people infected with HIV and, specifically, in those who receive episodic ART.

DETAILED DESCRIPTION:
HIV is a virus that can lead to AIDS, a disease that breaks down the immune system and allows for entry of life-threatening secondary infections. HIV is transmitted through the exchange of bodily fluids, primarily through sexual intercourse. Using ART treatments, people with HIV have been able to delay HIV replication and immune system deterioration and to improve quality of life. Data from the Strategies for Management of Antiretroviral Therapy (SMART) study indicate that episodic use of ART is associated with a higher risk of CVD than is continuous use of ART. The reasons behind this increased risk of CVD in the presence of HIV are not well understood. This study will determine mechanisms underlying the increased CVD risk among people infected with HIV and, specifically, in those who receive episodic ART.

This ancillary study to SMART will use relevant data and specimens from three subsamples of SMART participants and key subgroups. The three subsamples include participants randomly assigned to episodic or continuous ART, participants who had no previous use of ART prior to study entry or had ceased ART within 6 months prior to study entry, and participants who had experienced a CVD event with two matched controls for each case. The subgroups will include episodic and continuous ART participants who were taking either a protease inhibitor (PI) or non-nucleoside reverse transcriptase inhibitor (NNRTI) at study entry.

This current study will use previously collected SMART data. Researchers will use data on CD4+ count and HIV-RNA levels from a prebaseline study visit and follow-up study visits that occurred at Months 1 and 2, then every 2 months for Year 1, and every 4 months thereafter during the SMART study. In addition, this study will use baseline and yearly data provided by SMART participants on CVD risk factors and treatment, including use of drug treatments for high blood pressure, diabetes history, cholesterol levels, smoking history, white blood cell count, and height and weight measurements. Last, using plasma specimens that were collected at baseline, the Month 1 follow-up, and the final follow-up, researchers will compare changes in lipoprotein particle size and numbers, as measured by nuclear magnetic resonance (NMR) spectroscopy, and changes in inflammatory and coagulation markers.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the SMART study
* CD4+ lymphocyte count greater than 350 cells/mm3

Exclusion Criteria:

* Presence of life-threatening diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will utilize patient data and specimens already collected from the previous parent study, SMART.
Sampling Method: Probability Sample
Enrollment: 5472 (Actual)
Dates: Start 2002-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change in lipoprotein particles size and number | Measured at baseline, Month 1 follow-up visit, and last follow-up visit
Change in inflammatory and coagulation markers | Measured at baseline, Month 1 follow-up visit, and last follow-up visit
Reasons for increased CVD risk among HIV-infected individuals | Measured at study treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Duprez, MD, PhD, Principal Investigator — University of Minnesota

REFERENCES:
- [Result] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; El-Sadr WM, Lundgren J, Neaton JD, Gordin F, Abrams D, Arduino RC, Babiker A, Burman W, Clumeck N, Cohen CJ, Cohn D, Cooper D, Darbyshire J, Emery S, Fatkenheuer G, Gazzard B, Grund B, Hoy J, Klingman K, Losso M, Markowitz N, Neuhaus J, Phillips A, Rappoport C. CD4+ count-guided interruption of antiretroviral treatment. N Engl J Med. 2006 Nov 30;355(22):2283-96. doi: 10.1056/NEJMoa062360. PMID 17135583